CLINICAL TRIAL: NCT06812299
Title: Migraine and Work-disability: How Treatment with Monoclonal Antibodies Against CGRP Pathway Could Reduce Work-related Burden Among Migraine Population.
Brief Title: Work-related Burden Changes, Quantified with HEADWORK, Among Individuals Treated with Migraine Preventive Therapies.
Status: Completed | Type: Observational
Sponsor: IRCCS National Neurological Institute "C. Mondino" Foundation (Other)
Collaborators: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other); Fondazione Policlinico Universitario Campus Bio-Medico (Other)
Responsible Party: Sponsor
Other Study IDs: HEADWORK
Record Dates: First submitted 2025-01-17; First posted 2025-02-06 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2025-02

CONDITIONS: Headache (Migraine)
Keywords: PROM; Headwork; migraine related burden; presenteeism; absenteeism; ictal burden; interictal burden; work related burden; burden of disease
MeSH Terms: conditions — Migraine Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- High frequency episodic or chronic migraine: Patients affected by high frequency episodic migraine or chronic migraine with or without aura according to ICHD-III criteria who received treatment with monoclonal antibodies directed against the CGRP pathway.

SUMMARY:
Migraine is one of the leading causes of disability worldwide among the population under 50. It's economic indirect burden is mostly determined by reduction of work productivity both by absenteeism and presenteeism. Migraine work related burden was usually underestimated by commonly used patients reported outcomes (PROMs), until the introduction of the HEADWORK questionnaire, evaluating working difficulties and the factors that negatively impact work-related tasks. The investigators aim to assess the influence of anti-CGRP monoclonal antibodies on migraine work-related burden by means of this specific PROM.

DETAILED DESCRIPTION:
Migraine attributed burden is a complex and multifaceted entity encompassing patients, families, and society repercussions. It is identified with both an ictal burden, the consequences of pain and associated symptoms on individuals functioning during the migraine attack itself, and interictal burden, namely the limitations experienced between the attacks.

The disease burden is also associated with direct and indirect economic repercussions. According to a recent study, indirect costs mainly related to reduced work productivity, seems especially relevant. Reduction of work productivity may be defined in terms of absenteeism, loss of paid workdays, and presenteeism. The latter condition refers to days of impaired working performance due to migraine, and it is responsible of higher indirect costs. Many factors play a role in the identification of presenteeism, both related to the disease itself and the working place, making it difficult to precisely quantify it.

Commonly used PROMs have several limitations, this is why a specific PROM, known as HEADWORK questionnaire, was created to assess work-related difficulties and impairment in migraine individuals. HEADWORK is a 17-item, two-scale questionnaire that evaluates working difficulties in general or specific skills (such as problems solving or starting new tasks), and the factors that negatively impact work-related tasks (such as noise and brightness of the workplace).

Monoclonal antibodies directed against the Calcitonin Gene Related Peptide pathway (mAbs) represent a new targeted migraine preventive treatment. A recent study assessed the impact of mAbs in working-age migraine individuals, showing that the drug costs are compensated by reductions in both absenteeism and presenteeism, starting within the first three months of mAbs treatment Primary outcome is to assess changes in HEADWORK questionnaire, reflecting work-related difficulties, across one year treatment with mAbs in a population of migraine individuals.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of migraine without aura, migraine with aura, or chronic migraine according to the 3rd edition of the International Classification of Headache Disorder (ICHD-III);
* Patients eligible for treatment with anti-CGRP mAbs according to AIFA prescribing rules (at least 8 migraine days per month in the last three months, MIgraine Disability ASsessment score ≥ 11, and previous failure due to lack of efficacy or tolerability of at least three preventive drugs, among β-blockers, tricyclic antidepressants, antiepileptics, and onabotulinum- toxin-A (this latter only for chronic migraine)).

Exclusion Criteria:

* Subjects with contraindications for use of anti-CGRP mAbs;
* Concomitant diagnosis of medical diseases and/or comorbidities that, in the Investigator's opinion, might interfere with study assessments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients suffering from episodic and chronic migraine and eligible for treatment with anti-CGRP mAbs according to AIFA prescribing rules enrolled in the outpatients clinic of IRCCS C.Besta (Milan), IRCCS Mondino Foundation (Pavia) and Campus Biomedico (Rome)
Sampling Method: Non-Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2024-10-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in HEADWORK part 1 across 12 months of mAbs treatment (continuous variable) | Baseline (T0) - three months of mAbs treatment (T3) - six months of mAbs treatment (T6) - nine months of mAbs treatment (T9) - twelve months of mAbs treatment (T12)
  Changes from baseline in HEADWORK part 1 (11 item addressing migraine impact on work-related difficulties in general or specific skills) across 12 months of mAbs treatment compared to pre-treatment (continuous variable)
Changes from baseline in HEADWORK part 2 across 12 months of mAbs treatment compared to pre-treatment (continuous variable) | Baseline (T0) - three months of mAbs treatment (T3) - six months of mAbs treatment (T6) - nine months of mAbs treatment (T9) - twelve months of mAbs treatment (T12)
  Changes from baseline in HEADWORK (6 items addressing the factors contributing to working difficulties, defined as negative impact on work tasks) across 12 months of mAbs treatment compared to pre-treatment (continuous variable)

SECONDARY OUTCOMES:
Differences in monthly headache days across 12 months of mAbs treatment compared to pre-treatment (continuous variable) | Baseline (T0) - three months of mAbs treatment (T3) - six months of mAbs treatment (T6) - nine months of mAbs treatment (T9) - twelve months of mAbs treatment (T12)
  To evaluate differences in monthly headache days across 12 months of mAbs treatment compared to pre-treatment (continuous variable)
Differences in the intake of acute drugs per month across 12 months of mAbs treatment compared to pre-treatment (continuous variable) | Baseline (T0) - three months of mAbs treatment (T3) - six months of mAbs treatment (T6) - nine months of mAbs treatment (T9) - twelve months of mAbs treatment (T12)
  To evaluate differences in the intake of acute drugs per month across 12 months of mAbs treatment compared to pre-treatment (continuous variable)
Percentage of responders among individuals who completed 12 months of mAbs treatment (continuous variable) | Baseline (T0) - twelve months of mAbs treatment (T12)
  To evaluate the percentage of responders among individuals who completed 12 months of mAbs treatment, identified as those individuals who achieved a reduction of monthly headache frequency between 50% and 75% compared to baseline (continuous variable)
Percentage of super-responders among individuals who completed 12 months of mAbs treatment (continuous variable) | Baseline (T0) - twelve months of mAbs treatment (T12)
  To evaluate the percentage of super-responders among individuals who completed 12 months of mAbs treatment, identified as those individuals who achieved a reduction of monthly headache frequency >=75% compared to baseline (continuous variable)
Percentage of non responders among individuals who completed 12 months of mAbs treatment (continuous variable) | Baseline (T0) - twelve months of mAbs treatment (T12)
  To evaluate the percentage of non responders among individuals who completed 12 months of mAbs treatment, identified as those individuals who achieved a reduction of monthly headache frequency <50% compared to baseline (continuous variable)
Differences in HEADWORK part 2 across 12 months of mAbs treatment compared to pre-treatment according to response rate (continuous variable) | Baseline (T0) - three months of mAbs treatment (T3) - six months of mAbs treatment (T6) - nine months of mAbs treatment (T9) - twelve months of mAbs treatment (T12)
  To evaluate the differences in HEADWORK part 2 across 12 months of mAbs treatment compared to pre-treatment in the non-responder, responder and super-responder group (continuous variable)
Differences in HEADWORK part 1 across 12 months of mAbs treatment compared to pre-treatment according to response rate (continuous variable) | Baseline (T0) - three months of mAbs treatment (T3) - six months of mAbs treatment (T6) - nine months of mAbs treatment (T9) - twelve months of mAbs treatment (T12)
  To evaluate the differences in HEADWORK part 1 across 12 months of mAbs treatment compared to pre-treatment in the non-responder, responder and super-responder group (continuous variable)

CONTACTS AND LOCATIONS:
Overall Officials: Licia Grazzi, Dr, Principal Investigator — Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta
Locations (3):
- Italy (3):
  - Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta, Milan, Italy
  - IRCSS Mondino Foundation, Pavia, Italy
  - Policlinico Universitario Campus Biomedico, Rome, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Lazaro-Hernandez C, Caronna E, Rosell-Mirmi J, Gallardo VJ, Alpuente A, Torres-Ferrus M, Pozo-Rosich P. Early and annual projected savings from anti-CGRP monoclonal antibodies in migraine prevention: a cost-benefit analysis in the working-age population. J Headache Pain. 2024 Feb 12;25(1):21. doi: 10.1186/s10194-024-01727-0. PMID 38347485
- [Background] Steiner TJ, Terwindt GM, Katsarava Z, Pozo-Rosich P, Gantenbein AR, Roche SL, Dell'Agnello G, Tassorelli C. Migraine-attributed burden, impact and disability, and migraine-impacted quality of life: Expert consensus on definitions from a Delphi process. Cephalalgia. 2022 Nov;42(13):1387-1396. doi: 10.1177/03331024221110102. Epub 2022 Jul 5. PMID 35791285
- [Background] Raggi A, Covelli V, Guastafierro E, Leonardi M, Scaratti C, Grazzi L, Bartolini M, Viticchi G, Cevoli S, Pierangeli G, Tedeschi G, Russo A, Barbanti P, Aurilia C, Lovati C, Giani L, Frediani F, Di Fiore P, Bono F, Rapisarda L, D'Amico D. Validation of a self-reported instrument to assess work-related difficulties in patients with migraine: the HEADWORK questionnaire. J Headache Pain. 2018 Sep 10;19(1):85. doi: 10.1186/s10194-018-0914-7. PMID 30203193
- [Background] D'Amico D, Grazzi L, Grignani E, Leonardi M, Sansone E, Raggi A; HEADWORK Study Group. HEADWORK Questionnaire: Why Do We Need a New Tool to Assess Work-Related Disability in Patients With Migraine? Headache. 2020 Feb;60(2):497-504. doi: 10.1111/head.13735. Epub 2020 Jan 13. PMID 31943176
- [Background] GBD 2019 Diseases and Injuries Collaborators. Global burden of 369 diseases and injuries in 204 countries and territories, 1990-2019: a systematic analysis for the Global Burden of Disease Study 2019. Lancet. 2020 Oct 17;396(10258):1204-1222. doi: 10.1016/S0140-6736(20)30925-9. PMID 33069326
- [Background] Steiner TJ, Stovner LJ, Jensen R, Uluduz D, Katsarava Z; Lifting The Burden: the Global Campaign against Headache. Migraine remains second among the world's causes of disability, and first among young women: findings from GBD2019. J Headache Pain. 2020 Dec 2;21(1):137. doi: 10.1186/s10194-020-01208-0. No abstract available. PMID 33267788